CLINICAL TRIAL: NCT04135443
Title: Mobile App Promoting Sexual Health for Young Black Men Who Have Sex With Men
Brief Title: Evaluation of 3T, a Sex-Positive HIV/STI Mobile App Intervention for Young Black Men Ages 14-19 Attracted to Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETR Associates (Other)
Collaborators: dfusion Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3T
Record Dates: First submitted 2019-10-20; First posted 2019-10-22 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: HIV/AIDS and Infections; Sexual Behavior; Health Knowledge, Attitudes, Practice
Keywords: Healthy relationships
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Sexual Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: This is a two arm randomized controlled trial. Upon completing a baseline survey participants will be randomized into the intervention or an attention control condition. After randomization, participants will be granted access to their assigned mobile app (3T app or a general health website).
Masking Description: Participants are randomly assigned to their condition without being made aware of their assigned condition as "attention control" or "intervention." Each condition accesses materials online.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3T Tune in! Turn on! Turn up! (Experimental): The intervention is a mobile app delivered sexual health promotion program designed specifically for young black men who have sex with men or who are attracted to men. The mobile app includes 36 interactive activities including resource maps, pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP) content, and an asynchronous communication forum. The app helps participants to become clearer about what they do/don't want to do sexually, to communicate their choices. It also focuses on ways to increase healthy relationships, enhance sexual experience if having sex while reducing HIV/STI risk.
  Interventions: Behavioral: 3T Tune in! Turn on! Turn up!
- General Health Website Materials (Active Comparator): The control intervention features a website containing seven health promotion materials in online pamphlet or poster formats focusing on mental health (2 pamphlets), nutrition (2 pamphlets), relationships (2 pamphlets) and COVID (1 poster).
  Interventions: Behavioral: General Health Materials Website

INTERVENTIONS:
Behavioral: 3T Tune in! Turn on! Turn up! — A sex positive multimedia interactive mobile app delivered HIV/STI intervention developed for use by YBMSM ages 14-19. The program employs a theory based approach to address essential knowledge, perceptions of risk, peer norms, attitudes and skill with two primary goals: (1) To reduce HIV/STI the program emphasizes partner reduction, avoidance of concurrent partners, condoms and HIV/STI tests; and (2) To improve sexual health and relationships.
  Arms: 3T Tune in! Turn on! Turn up!
Behavioral: General Health Materials Website — The control group will receive access to a website containing general health promotion materials.
  Arms: General Health Website Materials

SUMMARY:
This study features a 2-arm randomized controlled trial with approximately 300 young black men who have sex with men (YBMSM) to assess the effectiveness of the 3T mobile app. To be eligible participants will be required to identify as male; Black, African-American, or biracial Black/African American; age 14-19 at baseline; self-identify as gay, bisexual, fluid, or sexually attracted to men; own a smartphone, and reside in any state in the United States. Those in the treatment arm will be provided with the 3T app and those in the control group will be given access to a website with general health materials. Participants will complete brief online surveys at baseline and at 3-months following the baseline to assess effectiveness in changing sexual risk behaviors and communication and condom use behaviors and attitudes.

DETAILED DESCRIPTION:
The overarching aim of this proposed Phase II research project is to fill a gap in prevention by completing the development and establishing the effectiveness of 3T: Tune in, Turn on, Turn up, a multimedia interactive sex-positive smartphone app-delivered HIV and other sexually transmitted infection (STI) intervention designed for use by YBMSM ages 14-19. The larger and longer term aims of developing an intervention specifically tailored to this population, utilizing a technology platform to reach youth where they are, is to contribute to a reduction in HIV/STI risk, increase HIV testing, and an increase in the quality of overall sexual health and relationships among YBMSM. To do this 3T emphasizes partner reduction, avoidance of concurrent partners, use of condoms if having anal or vaginal sex, and getting HIV/STI tests. 3T also focuses on improving quality of sexual experience and relationships, helping participants become clearer about what they do/don't want to do sexually, communicating their choices, and learning ways to enhance sexual experience without increasing HIV/STI risk. dfusion and its research partner, ETR, will meet the following specific Phase II aims:

* In conjunction with advisory panel members, develop content and corresponding storyboards for all activities. The curriculum will include content on risk reduction, sexual health and the quality of sexual experiences, and developing healthy relationships;
* Successful development of the first mobile app-delivered STI/HIV prevention program specifically designed for YBMSM aged 14-19. Reaching this aim requires continued development of the app technology, including the multimedia interactive activities, games, data collection, activity randomization, and an asynchronous forum. Research shows that YBMSM use the Internet to find information related to sex and sexuality, find friends and sexual partners, and YBMSM are increasingly using mobile apps, such as Grindr, to meet sex partners.20 The reliance on mobile devices for education and entertainment make it the ideal technology platform for reaching the YBMSM audience;
* Conduct a rigorous evaluation to determine the effectiveness of the intervention to reduce HIV/STI risk.

The evaluation features a 2-arm randomized controlled trial with approximately 300 young black men who have sex with men (YBMSM) to assess the effectiveness of the 3T mobile app. To be eligible participants will be required to identify as male; Black, African-American, or biracial Black/African American; age 14-19 at baseline; self-identify as gay, bisexual, fluid, or sexually attracted to men; own a smartphone, and reside in any state in the United States. Those in the treatment arm will be provided with the 3T app and those in the control arm will be asked to use a website with general health information. Participants will complete brief online surveys at baseline and at 3-months following the baseline to assess effectiveness in changing sexual risk behaviors and relationship and communication behaviors and attitudes.

Recruitment. We will use multiple methods to recruit participants: 1) Engaging Organizations. Approximately 15-20 organizations from across the U.S. that serve YBMSM will be approached to help recruit participants through social media and in-person 2) Using Social Media Advertising including targeted advertising on social media sites and sponsoring study posts with social media influencers in the YBMSM community.

ELIGIBILITY:
Inclusion Criteria:

1. self-identification of being aged 14-19;
2. ownership of an iphone or Android smartphone
3. self-identification of racial identity as black, African American, or biracial; and
4. self-identifying as gay, bisexual, same gender loving, or sexually attracted to the same gender.
5. capacity to assent, based on formal assessment
6. a willingness to participate after complete understanding of the topics of study, as indicated by a completed assent form
7. resides in the US

Exclusion Criteria:

* Anyone not meeting inclusion criteria

Ages: 14 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — self-identifying as gay, bisexual, same gender loving, or sexually attracted to the same gender
Enrollment: 178 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Kuhn, MS, Principal Investigator — dfusion Inc
Locations (1):
- ETR Associates, Scotts Valley, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 3T Tune in! Turn on! Turn up!: The mobile app includes 36 interactive activities including resource maps, pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP) content, and an asynchronous communication forum. Participants were randomly assigned individually to arms.
- General Health Website Materials: The control intervention featured a website containing seven health promotion materials in online pamphlet or poster formats focusing on mental health (2 pamphlets), nutrition (2 pamphlets), relationships (2 pamphlets) and COVID (1 poster). Participants were randomly assigned individually to study arms.
Period: Overall Study
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials
Started | 89 | 89
Completed | 74 | 74
Not Completed | 15 | 15

BASELINE CHARACTERISTICS:
Population: Young Black men who are attracted to men.
Groups:
- 3T Tune in! Turn on! Turn up!: The mobile app includes 36 interactive activities including resource maps, pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP) content, and an asynchronous communication forum.
- General Health Website Materials: The control intervention featured a website containing seven health promotion materials in online pamphlet or poster formats focusing on mental health (2 pamphlets), nutrition (2 pamphlets), relationships (2 pamphlets) and COVID (1 poster).
- Total: Total of all reporting groups
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials | Total
Number analyzed (Participants) | 89 | 89 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 18.28 (1.18) | 18.20 (1.25) | 18.23 (1.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 89 | 89 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 89 | 89 | 178
Engaged in condomless receptive or insertive anal or condomless vaginal intercourse last 3 months [Count of Participants; unit: Participants] | 57 | 54 | 111

OUTCOME MEASURES:

1. Primary Outcome: Condomless Anal Intercourse or Condomless Vaginal Intercourse
Description: Engaged in condomless receptive or insertive anal intercourse or condomless vaginal intercourse in the last 3 months
Time Frame: 3-months post baseline
Population: All participants with complete data on baseline and follow-up survey.
Measure: Count of Participants; unit: Participants
Groups:
- 3T Tune in! Turn on! Turn up!: The intervention is a mobile app delivered sexual health promotion program designed specifically for young black men who have sex with men or who are attracted to men. The mobile app includes 36 interactive activities including resource maps, pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP) content, and an asynchronous communication forum.
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials
Number analyzed (Participants) | 74 | 74
Participants | 49 | 50
Statistical Analysis 1: Comparison: 3T Tune in! Turn on! Turn up! vs General Health Website Materials; Test type: Superiority; p = 0.94, Regression, Logistic; Odds Ratio (OR) = 1.027, 95% CI 2-sided [0.511 to 2.063]

2. Secondary Outcome: Sexual Partners, no Condom, in the Last 3 Months
Description: # partners with whom had anal or vaginal sex without using condoms in the last 3 months
Time Frame: 3-months post baseline
Reporting Status: Not Posted

3. Secondary Outcome: Self-reported STI/HIV Testing in Last Three Months
Description: Number of times reported having been tested for STI, including HIV in the last 3 months
Time Frame: 3-months post baseline
Population: Participants with complete data on baseline and follow-up for outcome.
Measure: Mean (Standard Deviation); unit: Times tested, self reported
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials
Number analyzed (Participants) | 49 | 47
Times tested, self reported | 1.04 (1.70) | 0.60 (1.36)
Statistical Analysis 1: Comparison: 3T Tune in! Turn on! Turn up! vs General Health Website Materials; Test type: Superiority; p = 0.455, Regression, Linear — Threshold set to p<0.05; See analysis plan for covariates screened into model; Slope = 0.064

4. Secondary Outcome: Dyadic Communication Scale
Description: Scale measures beliefs regarding communication with partner about sexual desires/behavior. Average of 6 items on a 5-point scale (1 to 5), with a range of 1 - 5, with a higher score indicating better outcomes
Time Frame: 3-months post baseline
Population: Participants with complete data on baseline and follow-up survey for outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials
Number analyzed (Participants) | 73 | 70
score on a scale | 3.22 (0.62) | 3.22 (0.45)
Statistical Analysis 1: Comparison: 3T Tune in! Turn on! Turn up! vs General Health Website Materials; Test type: Superiority; p = 0.702, Regression, Linear — Threshold set to p<0.05; See analysis plan for covariates screened into model; Slope = 0.026

5. Secondary Outcome: Condom Attitudes Scale
Description: Scale measures attitudes regarding condoms. Average of 21 items on a 4-point scale (1 to 4), with a range of 1 - 4, with a higher score indicating better outcomes
Time Frame: 3-months post baseline
Population: Participants with complete baseline and follow-up survey data for outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials
Number analyzed (Participants) | 69 | 68
score on a scale | 3.02 (0.50) | 2.90 (0.44)
Statistical Analysis 1: Comparison: 3T Tune in! Turn on! Turn up! vs General Health Website Materials; Test type: Superiority; p = 0.375, Regression, Linear — Threshold set to p<0.05; See analysis plan for covariates screened into model; Slope = 0.049

6. Secondary Outcome: Condom Self-Efficacy Scale
Description: Scale measures perceived self-efficacy to use condoms. Average of 4 items on a 4-point scale (1 to 4), with a range of 1 - 4, with a higher score indicating better outcomes
Time Frame: 3-months post baseline
Population: Participants with complete data on baseline and follow-up survey for outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials
Number analyzed (Participants) | 70 | 67
score on a scale | 3.21 (0.69) | 3.07 (0.74)
Statistical Analysis 1: Comparison: 3T Tune in! Turn on! Turn up! vs General Health Website Materials; Test type: Superiority; p = 0.313, Regression, Linear — Threshold set to p<0.05; See analysis plan for covariates screened into model; Slope = 0.076

7. Secondary Outcome: Attitudes Towards Lube
Description: Scale measures attitudes towards lube. Average of 3 items on a 4-point scale (1-4), with a range of 1-4, with a higher score indicating more positive attitudes towards lube
Time Frame: 3-months post baseline
Population: Participants with complete data on baseline and follow-up survey for outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials
Number analyzed (Participants) | 72 | 69
score on a scale | 3.40 (0.63) | 3.40 (0.60)
Statistical Analysis 1: Comparison: 3T Tune in! Turn on! Turn up! vs General Health Website Materials; Test type: Superiority; p = 0.890, Regression, Linear — Threshold set to p<0.05; See analysis plan for covariates screened into model; Slope = -0.010

ADVERSE EVENTS:
Time Frame: Entire study period (Consent through 3 month follow-up), approximately 4 months.
Description: Used clinicaltrials.gov definitions.
Arm/Group | 3T Tune in! Turn on! Turn up! | General Health Website Materials
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/89
Other Adverse Events (participants affected / at risk) | 0/89 | 0/89

LIMITATIONS AND CAVEATS:
Small sample size limits generalizability; one short-term follow-up (3-month) survey limits insights on impacts; limited app use likely linked to lack of treatment effects, and the study lacked sufficient data to better understand all factors contributing to limits in app use; COVID impacted planned study recruitment and timeline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT04135443/Prot_SAP_000.pdf